CLINICAL TRIAL: NCT02109796
Title: a Controlled, Randomized Study Evaluating the Immediate Effect of One tDCS Session on Quadriceps Strength in Hemiparetic Patients.
Brief Title: Effects of tDCS on Quadriceps Strength After Stroke
Acronym: tDCS(HE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A00219-38
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Stroke
Keywords: tDCS; Stroke; Force; Spasticity; Gait; EMG; Isokinetic
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hemiplegic patient (Experimental): anodal transcranial direct current stimulation
  Interventions: Device: transcranial Direct current stimulation
- patient control (Sham Comparator): Sham transcranial direct current stimulation
  Interventions: Device: transcranial Direct current stimulation

INTERVENTIONS:
Device: transcranial Direct current stimulation

SUMMARY:
Previous studies show that one session of tDCS allow to improve muscle strength in hemiparetic patients in anodal condition. We test a new electrods configuration : a anodale stimulation opposite to the cortical representation area of the injured hemisphere and a simultaneous stimulation opposite to the homonyme the cortical representation area of the healthy hemisphere. This approach seems to be the best relevant electrods configuration in order to restore the inter-hemispheric balance.

We hypothesis that one session of tDCS with this electrods configuration allow to improve paretic quadriceps strength in hemiparetic patients after stroke.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* hemiparetic patient after stroke in chronic phase (> 6 months)
* capacity to walk with or without technical assistance
* following rehabilitation program for lower limbs

Exclusion Criteria:

* patient with bilateral brain lesion, cerebellar syndrom, and apraxia and/or aphasia
* previous orthopedic surgery in paretic lower limb (<6 moths)
* usual tDCS contraindications
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
maximum voluntary isometric strength of knee extensors | 2 hours
  The maximum voluntary isometric strength of paretic knee extensors will be evaluated with a isokinetic dynamometer, which measure peak torque.

SECONDARY OUTCOMES:
Resistive peak torque during passive knee flexion | 2h
Angle related to the resistive peak torque generation of the knee extensors | 2h
Amplitude of the interpolation twitch | 2h
EMG activation of the knee flexors and extensors during the strength evaluations (active and passive) | 2h
Functional evaluation of the gait performance and balance | 2h

CONTACTS AND LOCATIONS:
Overall Officials: Roche Nicolas, MD PH, Principal Investigator — Raymond Poincaré Hospital; Bensmail Djamel, MD PH, Principal Investigator — Raymond Poincare Hospital
Locations (1):
- Raymond Poincare Hospital, Garches, France

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411